CLINICAL TRIAL: NCT05745441
Title: Dinner Time for Obesity and Prediabetes
Acronym: DTOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00301239; K23DK133690 (NIH)
Record Dates: First submitted 2023-02-08; First posted 2023-02-27 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: PreDiabetes; Obesity; Healthy
Keywords: circadian; sleep; glucose; metabolism
MeSH Terms: conditions — Prediabetic State; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Dinner First (Experimental): Participants will be served dinner and a stable isotope of oral [2H31] palmitate to measure fat oxidation, at an early dinner time (before DLMO). This arm will then cross-over to Late Dinner as the second metabolic visit.
  Interventions: Behavioral: Early Dinner; Behavioral: Late Dinner; Drug: Early Dinner tracer; Drug: Late Dinner tracer
- Late Dinner First (Experimental): Participants will be served dinner and a stable isotope of oral [2H31] palmitate to measure fat oxidation, at a late dinner time (after DLMO). This arm will then cross-over to Early Dinner as the second metabolic visit.
  Interventions: Behavioral: Early Dinner; Behavioral: Late Dinner; Drug: Early Dinner tracer; Drug: Late Dinner tracer

INTERVENTIONS:
Behavioral: Early Dinner — Dinner before DLMO
Behavioral: Late Dinner — Dinner after DLMO
Drug: Early Dinner tracer — Stable isotope of oral [2H31] palmitate to measure fat oxidation, given with dinner before DLMO
Drug: Late Dinner tracer — Stable isotope of oral [2H31] palmitate to measure fat oxidation, given with dinner after DLMO

SUMMARY:
Obesity and its metabolic complications are leading causes of global morbidity and mortality. Evidence is mounting that inappropriate timing of food intake contributes to obesity. Specifically, late eating is associated with greater weight gain and metabolic syndrome. However, the mechanism by which late eating harms metabolism is not fully understood but may be related to mis-timing of food intake in relation to the body's endogenous circadian rhythm. Conversely, harmonization of eating timing with endogenous circadian rhythm may optimize metabolic health. In this study the investigators will use gold-standard methods of characterizing circadian rhythm in humans to examine the metabolic impacts food timing relative to endogenous circadian rhythm.

DETAILED DESCRIPTION:
This is a randomized, cross-over study that examines the metabolic impact of early vs late dinner, as defined by proximity of food intake to an individual's biological night as determined by dim light melatonin onset (DLMO) in normal-weight, healthy adult volunteers and in adults with obesity and prediabetes. Each participant will first undergo circadian phenotyping at the Johns Hopkins Bayview Clinical Research Unit (Baltimore, Maryland), with assessment of DLMO and core body temperature profile, as well as wrist actigraphy. Thereafter, participants will be crossover randomized to (1) a 24-hour metabolic chamber protocol where dinner is eaten 3 hours before DLMO (early dinner), or (2) a 24-hour metabolic chamber protocol where dinner is 1 hour eaten after DLMO (late dinner), both to be performed at the NIH Metabolic Clinical Research Unit (Bethesda, Maryland). The timing and nutritional contents of all meals, as well as sleep timing and duration, will be held constant. Oral [2H31] palmitate will be given with each dinner condition to quantify dietary fat oxidation. The 2 dinner conditions will occur in random order, with a 3- to 4-week washout period.

The investigators are enrolling both Normal-Weight Healthy (NWH) and Obesity-Prediabetes (OPD) research participants. At this time (5/2023) the investigators are focusing on the NWH group.

ELIGIBILITY:
The investigators are enrolling both Normal-Weight Healthy (NWH) and Obesity-Prediabetes (OPD) research participants. At this time (5/2023) the investigators are focusing on the NWH group.

Inclusion Criteria:

* For the Normal-Weight Healthy (NWH) cohort: Healthy male and female adults, age 18-50, with BMI 18-24.9 kg/m2 inclusively
* For the Obesity-Prediabetes (OPD) cohort: Male and female adults, age 18-50, with BMI ≥30 kg/m2 and prediabetes
* All participants must be able to understand study procedures, to comply with the procedures for the entire length of the study and be fully mobile.

Exclusion Criteria:

* Sleep disorder including insomnia, untreated moderate-severe sleep apnea, restless leg syndrome, or narcolepsy
* Night shift work
* Extreme delayed sleep phase defined as self-reported routine bedtime later than 1:00 AM or having mid-sleep on free days later than 5:00 AM on the Munich Chronotype Questionnaire (MCTQ) or DLMO later than 24:00
* Gastroesophageal reflux disease that affects ability to tolerate a dinner close to bedtime
* Active smoking
* Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Diabetes (type 1 or 2) or on any diabetes medications besides metformin
* Evidence of metabolic or cardiovascular disease, or disease that may influence metabolism (e.g. cancer, thyroid disease)
* Hemoglobin A1c ≥5.7% for NWH cohort; Hemoglobin A1c ≥6.5% for OPD cohort
* Hemoglobin < 10 g/dL
* Self-reported kidney disease
* Any known history of an inherited metabolic disorder
* Pregnant or lactating female (pregnancy test will be required prior to metabolic visits)
* Peri-menopausal or post-menopausal female as determined by follicle stimulating hormone of > 30 mIU/mL or fewer than 3 menstrual periods in 6 months
* Professional or collegiate athlete
* Participants who have travelled across time zones must have adequate time to recover from jet lag prior to enrollment (i.e., at least 3 days per time zone). Travel across >1 time zone after enrollment in the study will not be permitted.
* Weight less than 40 kg or more than 180 kg
* Gastrointestinal disorders that can lead to obstruction of the digestive tract (i.e. diverticular disease, history of bowel obstruction, inflammatory bowel disease, motility disorder)
* History of any surgical procedures in the gastrointestinal tract.
* Swallowing disorders
* Taking any prescription medication or other drug that may influence metabolism (e.g. diet/weight-loss medication, asthma medication, blood pressure medication, psychiatric medications, corticosteroids, or other medications at the discretion of the PI and/or study team)
* Chronic use of sedative hypnotics, anxiolytics, opiates
* Use of medications that can affect circadian rhythm (beta blockers, melatonin)
* Presence of a cardiac pacemaker or other implanted electro-medical devices
* Those who have to undergo strong electromagnetic field during the period of use of the ingestible thermosensor (i.e. MRI)
* Weight loss or gain of ≥ 5% of total body weight over the preceding 3 months
* Currently participating in a weight loss program
* Prior bariatric surgery
* Volunteers with strict dietary concerns (e.g. vegetarian or kosher diet, food allergies)
* History of significant intravenous access issues
* Non-English speaking individuals: The complexity of the instructions for various components of the study would make the study procedures difficult to follow in the setting of a language barrier.
* Other conditions or situations at the discretion of the PI

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
24-hour total fat oxidation | baseline, 4 weeks
  Within-subject difference in total fat oxidation between early dinner and late dinner conditions.

SECONDARY OUTCOMES:
4-hour post-prandial area-under-the-curve (AUC) glucose levels | baseline, 4 weeks
  Within-subject difference in post-prandial AUC glucose levels between early dinner and late dinner conditions.
4-hour post-prandial area-under-the-curve insulin levels | baseline, 4 weeks
  Within-subject difference in post-prandial AUC insulin levels between early dinner and late dinner conditions.
14-hour post-dinner cumulative dietary fat oxidation | baseline, 4 weeks
  Within-subject difference in dietary fat oxidation between early dinner and late dinner conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Jun, MD, Principal Investigator — Johns Hopkins University; Stephanie T Chung, MBBS, Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Yes
The investigators will provide raw data (without identifying information) to journals or other researchers upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be provided upon request within 1 year after publication and will be available to indefinitely.
Access Criteria: The PI will accept requests from other researchers who are examining pertinent outcomes.

REFERENCES:
- [Background] Gu C, Brereton N, Schweitzer A, Cotter M, Duan D, Borsheim E, Wolfe RR, Pham LV, Polotsky VY, Jun JC. Metabolic Effects of Late Dinner in Healthy Volunteers-A Randomized Crossover Clinical Trial. J Clin Endocrinol Metab. 2020 Aug 1;105(8):2789-802. doi: 10.1210/clinem/dgaa354. PMID 32525525
- [Background] Duan D, Gu C, Polotsky VY, Jun JC, Pham LV. Effects of Dinner Timing on Sleep Stage Distribution and EEG Power Spectrum in Healthy Volunteers. Nat Sci Sleep. 2021 May 14;13:601-612. doi: 10.2147/NSS.S301113. eCollection 2021. PMID 34017207
- See also: Screening Survey for DTOP — https://mrprcbcw.hosts.jhmi.edu/redcap/surveys/?s=LNACF9KWWDCCRXJ9